CLINICAL TRIAL: NCT00979134
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD4547 in Patients With Advanced Solid Malignancies
Brief Title: Study is Designed to Assess the Safety and Tolerability of AZD4547 at Increasing Doses in Patients With Advanced Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of study enrolment to Part C, Cohort 3 (08 July 2013) was based on the analysis of data from Study D2610C00004.
  Data were available from 33 patient
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2610C00001
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Cancer; Advanced Solid Malignancies
Keywords: Cancer; Tumour; Advanced Solid Malignancies; FGFR; Squamous NSCLC; Gastric adenocarcinoma
MeSH Terms: conditions — Neoplasms | interventions — AZD4547

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Experimental): Ascending doses of AZD4547 administered orally to patients to define the maximum tolerated dose (MTD) and/or a continuous, tolerable Recommended Dose (RD)
  Interventions: Drug: AZD4547
- Part B (Experimental): Dose expansion phase, at the RD defined in Part A
  Interventions: Drug: AZD4547
- Part C (Experimental): Expansion phase in patients with FGFR1 and FGFR2 amplified tumours commencing at the RD defined from Part A
  Interventions: Drug: AZD4547

INTERVENTIONS:
Drug: AZD4547 — Single dose is followed by washout 5-10 days before multiple dose, and at dose of 80mg twice daily
  Arms: Part B
Drug: AZD4547 — Patients start at a dose of 80 mg twice daily, with no washout
  Arms: Part C
Drug: AZD4547 — Single dose is followed by washout 5-10 days before multiple dose
  Arms: Part A

SUMMARY:
This study is primarily designed to assess the safety and tolerability of AZD4547 at increasing doses in patients with advanced solid malignancies and for whom no standard medication options are available. It also assesses the blood levels and action of AZD4547 in the body over a period of time.

ELIGIBILITY:
Inclusion Criteria:

* Minimum life expectancy of 12 weeks
* The presence of a solid, malignant tumour that is resistance to standard therapies or for which no standard therapies exist
* In the expansion for the study patients must have a tumour at least 1cm in size that can be measure using a CT or MRI scan, and provide a tumour sample to the sponsor company for testing of FGFR1 and/or 2 amplification
* Expansion, 5 groups of advanced cancer
* Solid tumours,FGFR1 and/or FGFR2 gene amplified
* Squamous NSCLC, FGFR1 gene low & high amplified
* Gastric adenocarcinoma, including the lower oesophagus/gastro-oesophageal junction, FGFR2 gene low & high amplified
* Aged at least 25 years

Exclusion Criteria:

* Treatment with any other chemotherapy, immunotherapy or anticancer agents within 3 weeks before the first dose of study
* An inability to be able to take the study medication
* A bad reaction to AZD4547 or any drugs similar to it in structure or class.

Ages: 25 Years to 149 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-10-21 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2015-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice André, Dr, Principal Investigator — Institut de cancérologie Gustave Roussy; Donal Landers, Dr, Study Director — AstraZeneca
Locations (27):
- United States (8):
  - Research Site, Stanford, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- France (2):
  - Research Site, Pierre-Bénite
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Cologne
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
- Italy (2):
  - Research Site, Napoli
  - Research Site, Rozzano
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
- Spain (3):
  - Research Site, Badajoz
  - Research Site, Majadahonda
  - Research Site, Valencia
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 21 October 2009 and last patient enrolled: 13 December 2013. This was a multicentre study conducted at a total of 29 centres in 7 countries.
Pre-assignment Details: In Parts A and B, a single dose was followed by a Washout Period of 5 to 10 days before multiple dosing commenced.
Groups:
- Part A: Dose escalation
- Part B: Dose expansion phase (80mg bd tablet)
- Part C: Dose expansion in patients with FGFR gene-amplified tumours
Period: Overall Study
Arm/Group | Part A | Part B | Part C
Started | 43 | 6 | 45
Completed | 10 (At DCO) | 0 (At DCO) | 5 (At DCO)
Not Completed | 33 | 6 | 40
Not completed — Disease progression | 18 | 2 | 5
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Death | 4 | 0 | 26
Not completed — Other | 8 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Part C (FISH Ratio >= 2); Part C (FISH Ratio < 2 ): Dose expansion in patients with FGFR gene-amplified tumours
- Total: Total of all reporting groups
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio < 2 ) | Part A | Total
Number analyzed (Participants) | 6 | 33 | 12 | 43 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (8.1) | 59.5 (10.82) | 58.2 (11.77) | 55.8 (10.1) | 57.59 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 16 | 3 | 18 | 40
  Male | 3 | 17 | 9 | 25 | 54

OUTCOME MEASURES:

1. Secondary Outcome: AUC(0-infinity)
Description: To characterise the pharmacokinetics (PK) of AZD4547 following a single administration and at steady state after dosing when given orally.
Time Frame: PK samples out to 96 hours "0 to 96 hours post-dose" after single dose (in parts A & B only). Steady state PK profile 3 weeks after the start of BD dosing.
Population: PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part C (FISH Ratio < 2): Dose expansion in patients with FGFR gene-amplified tumours
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio < 2) | Part A
Number analyzed (Participants) | 6 | 0 | 0 | 42
ng*h/mL | 1818 (59.43) |  |  | 2697 (110.8)

2. Secondary Outcome: Tumour Response (Best Objective Response) - Number of Patients With a Confirmed Response of Partial Response (PR) or Confirmed Response (CR)
Description: To obtain a preliminary assessment of the anti tumour activity of AZD4547 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) criteria version 1.1. Objective response = CR + PR; CR=disappearance of all target lesions and PR is >=30% reduction in sum of longest diameter of target lesions
Time Frame: Baseline assessment, then assessment every 6 weeks after start of treatment until objective disease progression.
Population: Efficacy/Tumour response: All dosed patients meeting the final FISH 6 score criteria with a baseline tumour assessment and had a FGFR1 FISH ratio ≥2 if the patient was from Part C
Measure: Number; unit: Patients
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part A | Part C (FISH Ratio < 2)
Number analyzed (Participants) | 6 | 33 | 43 | 12
Patients | 0 | 1 | 0 | 0

3. Secondary Outcome: Cmax (ng/mL)
Description: as for outcome 1
Time Frame: PK samples out to 96 hours "0-96 hours post dose" after single dose (in parts A & B only). Steady state PK profile 3 weeks after the start of BD dosing.
Population: PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part A | Part C (FISH Ratio < 2)
Number analyzed (Participants) | 6 | 0 | 43 | 0
ng/mL | 112.0 (81.47) |  | 167.4 (112.1) |

4. Secondary Outcome: Css,Max (ng/mL)
Description: as for outcome 1
Time Frame: PK samples out to 96 hours "0-96 hours post-dose" after single dose (in parts A & B only). Steady state PK profile 3 weeks after the start of BD dosing.
Population: PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part A | Part C (FISH Ratio < 2)
Number analyzed (Participants) | 6 | 0 | 32 | 0
ng/mL | 289.3 (45.98) |  | 297.1 (123.5) |

5. Secondary Outcome: AUC,ss(0-infinity)
Description: as for outcome 1
Time Frame: as for outcome 3
Population: PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio < 2) | Part A
Number analyzed (Participants) | 4 | 0 | 0 | 31
ng*h/mL | 2606 (41.32) |  |  | 2337 (125.2)

6. Primary Outcome: Number of Patients Who Experienced at Least 1 AE
Description: To investigate the safety and tolerability of AZD4547. System organ class (SOC), preferred term (PT), duration and severity all recorded.
Time Frame: AEs are monitored from screenng through to 30 day follow up period
Measure: Number; unit: Participants
Groups:
- Part C (FISH Ratio <2): Dose expansion in patients with FGFR gene-amplified tumours
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Participants | 6 | 33 | 12 | 43

7. Primary Outcome: Number of Participants Who Experienced at Least 1 Causally Related AE.
Description: To investigate the safety and tolerability of AZD4547. A causally related AE is an AE deemed to be causally related to AZD4547.
Time Frame: AEs are continually assessed from screening up to 30 day FU period
Measure: Number; unit: Participants
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Participants | 6 | 31 | 10 | 42

8. Primary Outcome: Number of Participants With at Least 1 AE of CTCAE >=G3
Description: To investigate the safety and tolerability of AZD4547
Time Frame: Ongoing up to discontinuation up to 30 day FU.
Measure: Number; unit: Participants
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Participants | 1 | 16 | 5 | 17

9. Primary Outcome: Number of Participants With at Least 1 Causally Related AE of CTCAE >=G3
Description: To investigate the safety and tolerability of AZD4547
Time Frame: Ongoing up to discontinuation up to 30 day FU.
Measure: Number; unit: Participants
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Participants | 0 | 8 | 3 | 12

10. Primary Outcome: Number of Participants Who Experienced at Least One SAE
Description: To investigate the safety and tolerability of AZD4547. A SAE (Serious Adverse Event) is and AE (adverse Event) which fulfills one of the following criteria that the PI assesses closely such as results in death, immediately life-threatening, requires hospitalisation or prolongation of, results in significant disability, results in birth defect, may jepardise the patient or require intervention to prevent any of the previous outcomes.
Time Frame: Serious Adverse Events (SAEs) are continually assessed from Screening up to the end of the 30 day FU period.
Measure: Number; unit: Number of participants
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Number of participants | 1 | 10 | 3 | 11

11. Primary Outcome: Number of Participants With at Least 1 Causally Related SAE
Description: To investigate the safety and tolerability of AZD4547: SAEs are assessed and deemed as causally related or not to AZD4547
Time Frame: SAEs are continually monitored from screening to end of 30 FU period
Measure: Number; unit: Number of participants
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio <2) | Part A
Number analyzed (Participants) | 6 | 33 | 12 | 43
Number of participants | 1 | 5 | 0 | 5

ADVERSE EVENTS:
Time Frame: AEs were collected on a continual basis from Screening up until the end of the 28 day follow up period.
Groups:
- Part C (FISH Ratio < 2): Dose expansionj in patients with FGFR gene-amplified tumours
Arm/Group | Part B | Part C (FISH Ratio >= 2) | Part C (FISH Ratio < 2) | Part A
Serious Adverse Events (participants affected / at risk) | 1/6 | 10/33 | 3/12 | 11/43
Other Adverse Events (participants affected / at risk) | 6/6 | 33/33 | 12/12 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B (N=6) | Part C (FISH Ratio >= 2) (N=33) | Part C (FISH Ratio < 2) (N=12) | Part A (N=43)
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
ALT increased (Investigations) | 0 | 0 | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 0 | 1 (1)
GGT increased (Investigations) | 0 | 0 | 0 | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 0 | 0 | 0 | 1 (1)
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 (1)
Tumour associated fever (General disorders) | 0 | 0 | 0 | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 2 (2) | 1 (1) | 0
Asthenia (General disorders) | 0 | 1 (1) | 1 (1) | 0
Chorioretinopathy (Eye disorders) | 0 | 2 (2) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 (2) | 0 | 0
Atrial flutter (Vascular disorders) | 0 | 0 | 1 (1) | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0
Decreased appetite (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 (1) | 0
Epilepsy (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Euthanasia (Social circumstances) | 0 | 1 (1) | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Hypotension (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Pericardial effusion (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 (1) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 (1) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part B (N=6) | Part C (FISH Ratio >= 2) (N=33) | Part C (FISH Ratio < 2) (N=12) | Part A (N=43)
Constipation (Gastrointestinal disorders) | 3 (3) | 13 (13) | 0 (0) | 24 (24)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (8) | 0 (0) | 21 (21)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 15 (15) | 0 (0) | 18 (18)
Stomatis (Gastrointestinal disorders) | 5 (5) | 10 (10) | 6 (6) | 18 (18)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 0 | 20 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (8) | 0 (0) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 12 (12) | 4 (4) | 14 (14)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 0 (0) | 15 (15)
Vomiting (Gastrointestinal disorders) | 3 (3) | 10 (10) | 5 (5) | 11 (11)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 11 (11) | 6 (6) | 12 (12)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9) | 0 (0) | 11 (11)
Fatigue (General disorders) | 2 (2) | 13 (13) | 4 (4) | 10 (10)
Asthenia (General disorders) | 2 (2) | 4 (4) | 0 (0) | 9 (9)
Dry eye (Eye disorders) | 0 | 9 (9) | 0 (0) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 0 (0) | 8 (8)
Headache (Nervous system disorders) | 2 (2) | 0 | 0 | 6 (6)
Pyrexia (General disorders) | 1 (1) | 0 | 0 | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 | 0 | 5 (5)
Dyspepsia (Nervous system disorders) | 1 (1) | 0 | 0 | 5 (5)
Muscle spasms (Nervous system disorders) | 1 (1) | 0 | 0 | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 | 0 | 4 (4)
Breath sounds abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 5 (5) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 13 (13)
Ageusia (Metabolism and nutrition disorders) | 4 (4) | 0 | 0 | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 10 (10)
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 7 (7)
Oedema peripheral (Eye disorders) | 0 | 0 | 0 | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 5 (5)
ALT increased (Investigations) | 0 | 0 | 0 | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 4 (4)
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 5 (5)

LIMITATIONS AND CAVEATS:
Due to early termination no AUC(inf), Cmax, Css,max and AUC,ss for Part C (PK). Data from 33 patients after 22 days of multiple dosing in Part A & limited data for part B only.

1 subject not dosed, so pre-stated subject number 95, total with data 94.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other